CLINICAL TRIAL: NCT05070338
Title: Reducing Inappropriate Prescription Opioid Prescribing at Hospital Discharge
Brief Title: Postoperative Nudges to Reduce Opioid Prescribing
Acronym: POST-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Sutter Health (Other); University of California, Los Angeles (Other); University of Southern California (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01DA046226 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-10-07 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Opioid Prescribing
Keywords: Opioid Epidemic; Inappropriate Prescribing; Opioid-Related Disorders; Practice Guideline; Peer Influence; Nudges
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guideline-Based Nudges (Experimental)
  Interventions: Behavioral: Guideline-Based (Injunctive Norm) Nudges
- Peer-Based Nudges (Experimental)
  Interventions: Behavioral: Peer-Based (Social Norm) Nudges
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Guideline-Based (Injunctive Norm) Nudges — Surgeons in this arm will receive an email with the following content at the end of each month in which at least two of their patients are discharged with an opioid prescription that exceeds the prescribing guideline for the procedure performed.
  Dear Dr. [Name],
  In [month], at least XX of your patients were discharged with opioid prescriptions exceeding the amounts recommended by safety guidelines for these procedures.
  For patient safety, Sutter Health recommends prescribing within the ranges below for these procedures. Doing so will also meet best-practice safety guidelines for post-operative opioid prescribing.
  We will continue to send you opioid prescribing safety reports.
  Sincerely, [Signature]
  [Table displaying recommended ranges of 5mg oxycodone tablets for each procedure]
  Arms: Guideline-Based Nudges
Behavioral: Peer-Based (Social Norm) Nudges — Surgeons in this arm will receive an email with the following content at the end of each month in which at least two of their patients are discharged with an opioid prescription that exceeds the prescribing guideline for the procedure performed.
  Dear Dr. [Name],
  In [month], at least XX of your patients were discharged with opioid prescriptions exceeding the amount prescribed by YY% of your peers for these procedures.
  YY% of [specialty] surgeons at Sutter Health prescribe within the ranges below for these procedures.
  We will continue to send you opioid prescribing safety reports.
  Sincerely, [Signature]
  [Table displaying recommended ranges of 5mg oxycodone tablets for each procedure]
  The ranges of 5mg oxycodone tablets displayed will be the same as the ranges stipulated by the prescribing guidelines, but this nudge will not mention guidelines.
  Arms: Peer-Based Nudges

SUMMARY:
This study tests the effectiveness of two email-based behavioral nudges, one based on peer behavior and one based on best practice guidelines, in reducing excessive opioid prescriptions after surgery. It will be conducted in three surgical specialties (general surgery, orthopedic surgery, and obstetric/gynecological surgery) at 19 hospitals within one healthcare system. These specialties will each be randomized to a control group or one of two nudge groups. Each month for one year, surgeons in the nudge groups will receive emails comparing their opioid prescribing either to their peers' prescribing or to prescribing guidelines. Both types of email-based nudges are expected to reduce opioid prescribing after surgery.

ELIGIBILITY:
The nudges that a surgeon in either intervention arm will receive are based on that surgeon's eligible discharge opioid prescriptions in the previous month. Eligible prescriptions meet all of the following criteria:

* the patient is at least 18 years old at the date of surgery
* the patient is discharged to their home
* the surgical procedure has an applicable post-operative opioid prescribing guideline
* the surgical procedure is the only surgical procedure performed during the patient's hospital stay
* the prescription is for an opioid taken orally (tablets, capsules, or liquid solution)

To avoid contamination between the intervention arms, surgeons who operate across multiple surgical specialties (defined as surgeons who performed less than 90% of their total procedures in one specialty between June 2020 and May 2021) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Watkins, MD, MSHS, Principal Investigator — RAND
Locations (1):
- Sutter Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon reasonable request.

REFERENCES:
- [Derived] Martinez MC, Bouskill K, Yan XS, Kirkegaard A, Doctor JN, Watkins KE. A qualitative analysis on the implementation of a nudge intervention to reduce post-surgical opioid prescribing. BMC Health Serv Res. 2025 Apr 8;25(1):512. doi: 10.1186/s12913-025-12651-7. PMID 40200214
- [Derived] Martinez M, Kirkegaard A, Bouskill K, Yan XS, Wagner Z, Watkins KE. Surgeons' views of peer comparison and guideline-based feedback on postsurgery opioid prescriptions: a qualitative investigation. BMJ Open Qual. 2024 Apr 5;13(2):e002750. doi: 10.1136/bmjoq-2024-002750. PMID 38580444
- [Derived] Wagner Z, Kirkegaard A, Mariano LT, Doctor JN, Yan X, Persell SD, Goldstein NJ, Fox CR, Brummett CM, Romanelli RJ, Bouskill K, Martinez M, Zanocco K, Meeker D, Mudiganti S, Waljee J, Watkins KE. Peer Comparison or Guideline-Based Feedback and Postsurgery Opioid Prescriptions: A Randomized Clinical Trial. JAMA Health Forum. 2024 Mar 1;5(3):e240077. doi: 10.1001/jamahealthforum.2024.0077. PMID 38488780
- [Derived] Kirkegaard A, Wagner Z, Mariano LT, Martinez MC, Yan XS, Romanelli RJ, Watkins KE. Evaluating the effectiveness of email-based nudges to reduce postoperative opioid prescribing: study protocol of a randomised controlled trial. BMJ Open. 2022 Sep 19;12(9):e061980. doi: 10.1136/bmjopen-2022-061980. PMID 36123066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: October 19, 2021; Primary Completion Date: October 18, 2022; Study completion date: October 18, 2023. Participants were recruited from hospitals in the Sutter care health system.
Units Other Than Participants: Specialty-hospital clusters
Groups:
- Control: No intervention
Period: Overall Study
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Started | 216; 19 Specialty-hospital clusters | 207; 19 Specialty-hospital clusters | 217; 19 Specialty-hospital clusters
Completed | 216; 19 Specialty-hospital clusters (Over the intervention year, the 216 surgeons in the Guideline-Based Nudges arm were responsible for 15459 patient discharges meeting the study eligibility criteria. The patients themselves were not enrolled in the study.) | 207; 19 Specialty-hospital clusters (Over the intervention year, the 207 surgeons in the Peer-Based Nudges arm were responsible for 10752 patient discharges meeting the study eligibility criteria. The patients themselves were not enrolled in the study.) | 217; 19 Specialty-hospital clusters (Over the intervention year, the 217 surgeons in the control arm were responsible for 12024 patient discharges meeting the study eligibility criteria. The patients themselves were not enrolled in the study.)
Not Completed | 0; 0 Specialty-hospital clusters | 0; 0 Specialty-hospital clusters | 0; 0 Specialty-hospital clusters

BASELINE CHARACTERISTICS:
Population: Surgeons in the Sutter Health hospital system
  Note: Only surgeons were enrolled in the study. Patients were not enrolled in the study and so their characteristics were not assessed at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control | Total
Number analyzed (Participants) | 216 | 207 | 217 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (17.6) | 50.1 (17.3) | 53.7 (17.7) | 51.3 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 87 | 87 | 257
  Male | 133 | 120 | 130 | 383
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Discharges With Opioid Prescriptions Above Prescribing Guidelines
Description: Prescriptions will be compared to prescribing guidelines via morphine milligram equivalents (MMEs) and coded as within or above guidelines. If no opioid is prescribed at discharge, this will be coded as within guidelines.
Time Frame: 12 months
Population: The units analyzed are the discharges of patients operated on by surgeons enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Proportion of discharges
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Proportion of discharges | 0.254 [0.247 to 0.261] | 0.275 [0.267 to 0.284] | 0.368 [0.359 to 0.376]

2. Secondary Outcome: Morphine Milligram Equivalents (MMEs) Prescribed at Discharge
Description: Continuous measure of the total morphine milligram equivalents prescribed at discharge
Time Frame: 12 months
Population: The units analyzed are the discharges of patients operated on by surgeons enrolled in the study.
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents (MMEs)
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Morphine milligram equivalents (MMEs) | 78.7 [76.8 to 80.6] | 58.6 [57.0 to 60.2] | 67.6 [65.9 to 69.3]

3. Secondary Outcome: Days' Supply of Opioids Prescribed at Discharge
Description: Continuous variable indicating the number of days' supply of opioids prescribed at discharge
Time Frame: 12 months
Population: Contrary to initial expectations, the days' supply of opioids prescribed at discharge was not captured by the Sutter Health electronic health records system. This outcome measure could therefore not be assessed.
  The quantity of opioids prescribed at discharge is still captured similarly by the outcome measure Morphine Milligram Equivalents (MMEs) Prescribed at Discharge.
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of Discharges Where Any Opioid Was Prescribed
Description: Derived from a binary variable indicating whether any opioid was prescribed at discharge
Time Frame: 12 months
Population: The units analyzed are the discharges of patients operated on by surgeons enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Proportion of discharges
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Proportion of discharges | 0.484 [0.476 to 0.491] | 0.476 [0.466 to 0.485] | 0.518 [0.509 to 0.527]

5. Secondary Outcome: Proportion of Patients on Opioids for Greater Than 3 Months Post-discharge
Description: Derived from a binary variable indicating whether the patient has any opioid prescriptions between 3 and 6 months after surgery
Time Frame: 3-6 months post-discharge
Population: The units analyzed are the discharges of patients operated on by surgeons enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Proportion of discharges
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Proportion of discharges | 0.123 [0.118 to 0.128] | 0.099 [0.093 to 0.105] | 0.102 [0.097 to 0.108]

6. Secondary Outcome: Number of 30-day All-cause Emergency Department Visits
Description: Number of emergency department visits the post-operative patient has in the 30 days after the initial procedure
Time Frame: 0-30 days post-discharge
Population: The units analyzed are the post-operative discharges of patients operated on by surgeons enrolled in the study. For patients who had multiple procedures in multiple admissions over the study period, each discharge is counted separately.
Measure: Mean (95% Confidence Interval); unit: Emergency department visits
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Emergency department visits | 0.062 [0.058 to 0.067] | 0.057 [0.052 to 0.062] | 0.062 [0.057 to 0.067]

7. Secondary Outcome: Number of 30-day All-cause Hospitalizations
Description: Number of hospital admissions the post-operative patient has in the 30 days after the initial procedure
Time Frame: 0-30 days post-discharge
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Hospital admissions
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Hospital admissions | 0.023 [0.021 to 0.026] | 0.029 [0.025 to 0.032] | 0.023 [0.020 to 0.026]

8. Secondary Outcome: Proportion of Discharge Opioid Prescriptions Above Prescribing Guidelines in the Year After the Intervention Ends
Description: as for outcome 1
Time Frame: 12 months (months 13-24 of the study)
Population: The units analyzed are the discharges of patients operated on by surgeons enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Proportion of discharges
Units Other Than Participants: Patient discharges
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
Number analyzed (Participants) | 216 | 207 | 217
Number analyzed (Patient discharges) | 15459 | 10752 | 12024
Proportion of discharges | 0.253 [0.246 to 0.261] | 0.250 [0.241 to 0.259] | 0.363 [0.354 to 0.372]

ADVERSE EVENTS:
Time Frame: 13 months
Description: A data and safety monitoring board monitored adverse events within 30 days of discharge among patients of enrolled surgeons. The numbers of participants at risk reported reflect the number of patient discharges. Surgeons were not monitored for adverse effects given the minimal risk of receiving emails.
  Only hospitalizations, ED visits, and opioid refills were monitored. Mortality was not monitored because the intervention did not pose a mortality risk.
Arm/Group | Guideline-Based Nudges | Peer-Based Nudges | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1096/15459 | 755/10752 | 849/12024
Other Adverse Events (participants affected / at risk) | 3045/15459 | 1752/10752 | 1617/12024
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guideline-Based Nudges (N=15459) | Peer-Based Nudges (N=10752) | Control (N=12024)
All-Cause Hospitalizations (General disorders) | 327 | 279 | 249
All-Cause Emergency Department Visits (General disorders) | 829 | 537 | 641
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guideline-Based Nudges (N=15459) | Peer-Based Nudges (N=10752) | Control (N=12024)
Opioid Refills (General disorders) | 3045 | 1752 | 1617

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT05070338/Prot_SAP_000.pdf